CLINICAL TRIAL: NCT04192045
Title: Quality of Recovery From Obstetric Anaesthesia - a Multicentre Study
Acronym: ObsQoR
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS254064
Record Dates: First submitted 2019-11-08; First posted 2019-12-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Obstetric Anesthesia Problems; Anesthesia Morbidity; Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be taken from selected Caesarean Delivery Patients before and after delivery to analyse to assess immune profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A survey will be used at 24 hours and 30 days to assess the quality of recovery

SUMMARY:
Quality of recovery is an important outcome measure in anaesthesia, whilst there are validated tools for this in surgery and regional anesthesia there are no fully validated tools for obstetrics anaesthesia. The aim of this study is to use the Obstetric Quality of Recovery (ObsQoR) score across multiple centres to assess correlation to length of stay and variation for different types of operative and non- operative delivery.

DETAILED DESCRIPTION:
An observational survey based study, for 3 consecutive week days, chosen by the local investigating team during a two-week period across multiple centres.

* Local investigators will complete the survey with each patient who has received anaesthetic intervention from an anaesthetist, 1 day, around 24hrs after delivery in line with their routine anaesthetic follow up.
* At 30 days, a telephone survey will be conducted with each patient to repeat the ObsQoR survey and ask key questions regarding functional recovery and activities of daily living post delivery.

In addition for a small number of sites, elective caesarean delivery patients will have blood taken at the point of anaesthesia and 24 hours post delivery to assess the immune function and any changes which may predict poorer outcome in these women.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients over 18 years old.
* Intervention occurring after 32/40 gestation.
* All mothers receiving anaesthesia or anaesthetic analgesia during their peripartum period.

Exclusion Criteria:

* Unable to comprehend the questions asked
* Patient refusal
* Under 32/40 weeks gestation
* Cervical cerclage insertion or removal, anaesthesia for External Cephalic Verison
* Neonatal death
* Non- NHS patients

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female peripartum
Study Population: Peripartum women during the designated study period who have received anaesthetic intervention in the previous 24-hour period for 3 consecutive days.
Sampling Method: Non-Probability Sample
Enrollment: 1638 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
• Correlation of ObsQoR with length of hospital stay (LOS) in hours following delivery across multiple centres, particularly ObsQoR score and prediction of prolonged LOS (>1.5 SD) and readmission to hospital. | Up to 3 months
  During the study the total length of stay in hours will be calculated for participating patients. This will be correlated with the score from the ObsQoR survey tool. In addition the readmission status of the patient will be asked at the subsequent survey combined with the patient's health care record to correlate with the ObsQoR tool score. Where the ObsQoR score is measured between 0-100 and LOS will be in hours. Readmission will be a binary outcome measure
• The relationship between ObsQoR and patient-reported ready for discharge. This will concurrently be determined to account for institutional, non-medical maternal factors neonatal factors that may delay discharge and impact LOS. | up to 3 months
  The patient will be surveyed using the ObsQoR tool and also asked regarding when they felt they were ready for discharge to take into account the multitude of factors which may impact on the overall length of stay. Where the ObsQoR score is measured between 0-100 and LOS will be in hours.

SECONDARY OUTCOMES:
• Comparing ObsQoR profiles with differing types of obstetric anaesthesia and delivery method. | up to 3 months
  ObsQoR tool will be used to assess the quality of recovery from General anaesthesia and differing types of regional anaesthesia (Spinal, Epidural, Dural puncture epidural (DPE) and combined spinal and epidural (CSE)
• Variations in ObsQoR scores across differing centres. | up to 3 months
  A multicentreed evaluation of the ObsQoR score across multiple centres
• Impact of patient factors on ObsQoR score. | up to 3 months
  A large number of variables will affect the quality of recovery and the ObsQoR score, these factors will be assessed. Where the ObsQoR score is measured between 0-100
• Impact of anaesthetic or obstetric factors on ObsQoR score. | up to 3 months
  A large number of variables will affect the quality of recovery and the ObsQoR score, these factors will be assessed. Where the ObsQoR score is measured between 0-100
• Impact of neonatal facts on ObsQoR score. | up to 3 months
  A large number of variables will affect the quality of recovery and the ObsQoR score, these factors will be assessed. Where the ObsQoR score is measured between 0-100
• Impact of institutional factors on ObsQoR score. | up to 3 months
  Differing centres will have differing institutional setup, guidelines, staffing levels, these will be assessed related to ObsQoR scores. Where the ObsQoR score is measured between 0-100
• Impact of time of day on ObsQoR score. | up to 3 months
  Time of day may impact on patient care on the quality of recover and the ObsQoR score- these will both be assessed. Where the ObsQoR score is measured between 0-100
• Impact of anaesthesia provider factors on ObsQoR score. | up to 3 months
  The level of seniority of anaesthesia provider may impact on the quality of recover and the ObsQoR score- these will both be assessed. Where the ObsQoR score is measured between 0-100
• Prediction of patients who are likely to have an ongoing requirement for analgesia. | up to 3 months
  The varying delivery methods have differing requirements for analgesia, it is not currently known the impact and effect this has on the quality of recovery. Where the ObsQoR score is measured between 0-100
• Prediction of patients who are likely to require further follow up in the community or investigation. | up to 3 months
  The patient surgical social and institutional demographics which may predispose some patients to seek healthcare in either the community or hospital setting
• Prediction of patients' ability to return to normal activities of daily living. | up to 3 months
  Functional recovery will be assessed observing return to normal activities of daily living (ADLs) and compared to ObsQoR score for patients of all delivery types. The score of ADLs will be correlated to ObsQoR score Where the ObsQoR score is measured between 0-100
• Prediction of patients' who are unable to achieve adequate activity levels. As determined by number of steps on mobile phone / activity tracker. | up to 3 months
  Assessment of the number of steps and related to quality of recovery and return to normal activities of daily living. Where steps will be a continuous measure and ObsQoR score will be measured from 0-100.
Assessment of perioperative immune function and response to surgical trauma as a predictor of outcome following elective caesarean delivery. | up to 3 months
  this will be assessed by taking bloods at the point of anaesthesia and 24 hours post in selected patients undergoing a elective caesarean delivery. The samples will then be analysed to assess the immune response.
Assessment of correlation between ObsQoR scores, EQ-5D and global health visual analogue scale results at 24 hours and 30 days. | up to 30 days
  Assessment of the relationship between ObsQoR scores at 24 hours with EQ-5D and global VAS scores at 24 hours and 30 days between different patients modes of anaesthesia, delivery types and institutions. Assessment of the relationship patient reported outcome measures PROMs to objective poor recovery such as, length of stay, complications and readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Kariem El-Boghdadly, Study Chair — GSTT
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The raw data will be available on request at the discretion of the central study team